CLINICAL TRIAL: NCT01254890
Title: Phase I/II Study of Sorafenib and 5-Azacitidine for the Treatment of Patients With Refractory or Relapsed Acute Leukemia and Myelodysplastic Syndrome (MDS) - (VZ-MDS-PI-0227)
Brief Title: Sorafenib and 5-Azacitidine in Acute Leukemia + Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry); Onyx Therapeutics, Inc. (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0511; NCI-2011-00257 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Results first posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-03

CONDITIONS: Leukemia
Keywords: Relapsed Acute Leukemia; Chronic Myelomonocytic Leukemia; CMML; Myelodysplastic Syndrome; MDS; Acute myeloid leukemia; AML; 5-azacitidine; Azacitidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Sorafenib; Nexavar; BAY43-9006
MeSH Terms: conditions — Leukemia; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacitidine + Sorafenib (Experimental): Azacitidine (AZA) 75 mg/m^2 subcutaneously (SQ) or intravenously (IV) daily for 7 days; Sorafenib 200 mg orally twice a day.
  Interventions: Drug: Azacitidine; Drug: Sorafenib

INTERVENTIONS:
Drug: Azacitidine — 75 mg/m^2 subcutaneously (SQ) or by vein (IV) daily for 7 days per 28 day cycle.
  Other Names: 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
Drug: Sorafenib — Starting dose level 200 mg by mouth two times a day in a 28 day cycle. In Phase II, Sorafenib administered per MTD dose from Phase I. Drug doses separated by approximately 12 hours.
  Other Names: Nexavar; BAY43-9006

SUMMARY:
The goal of this clinical research study is to learn if 5-azacitidine and sorafenib can control the disease in patients with AML or MDS. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Sorafenib is designed to block the function of important proteins in cancer cells. These proteins, when active, are partly responsible for the abnormal growth and behavior of cancer cells.

5-Azacytidine is designed to activate ("turn on") certain genes in cancer cells whose job is to fight tumors.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive 5-azacytidine either under the skin or by vein on Days 1-7 of each 28-day cycle. If by vein, the infusion will take about 10-40 minutes.

You will take sorafenib by mouth 2 times a day about 12 hours apart, with water on empty stomach, every day.

Each study cycle may last a little longer than 28 days, depending on how you are doing.

Study Visits:

Every week, blood (about 1 tablespoon) will be drawn for routine tests.

Every week for the first 6 weeks, and then as often as your doctor thinks it is needed, you will have your blood pressure measured.

Before each cycle:

* Your performance status will be recorded.
* You will have a physical exam, including measurement of your blood pressure and weight.

Before every 2-4 cycles, you will have a bone marrow aspirate to check the status of the disease.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse or intolerable side effects occur.

Your participation on the study will be over once you have completed the end-of-treatment and follow-up visits.

End of Study Drug Administration Visit:

After you have stopped taking the study drugs, the following tests and procedures will be performed:

* Your medical history will be recorded.
* Your performance status will be recorded.
* You will have a physical exam, including measurement of your blood pressure and weight.
* You will have a bone marrow aspirate collected to check the status of disease.

This is an investigational study. Sorafenib is FDA approved and commercially available for kidney cancer and liver cancer. 5-Azacitidine is FDA approved for the treatment of MDS, but its combination with sorafenib is investigational.

Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MDS, CMML or AML, who have failed pror therapy (including low and intermediate risk patient who have required prior therapy).
2. Patients with MDS or CMML should have failed prior therapy with a hypomethylating agent and/or with lenalidomide. Patients who have received prior azacitidine are eligible if the treating physician feels that participation in the sudy is in the patients' best interest.
3. Patients with AML should have failed any prior induction therapy or have relapsed after prior therapy.
4. Patients with MDS or CMML who received therapy with hypomethylating agent and progress to AML are eligible at the time of diagnosis of AML regardless of any prior therapy for AML.
5. Patients with any of the eligible diagnoses who have received no prior therapy are eligible if not candidates to receive or refuse standard therapy.
6. Age of greater than or equal to 18 years of age.
7. ECOG Performance Status less than or equal to 2.
8. Adequate liver (bilirubin less than or equal 1.5 * upper limit of normal (ULN), ALT and AST less than or equal 2.5 * ULN and Alkaline phosphatase less than 4 * ULN if not related to leukemic disease) and renal (creatinine less than or equal 1.5* ULN) function. Amylase and Lipase must be less than or equal 2 * ULN.
9. Patients must provide written informed consent.
10. Patients must have been off chemotherapy for 2 weeks prior to entering this study, unless there is evidence of rapidly progressive disease, and must have recovered from the toxic effects of that therapy to at least grade 1. Use of hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy but should be stopped for 24 hours prior to initiation of azacitidine.
11. Women of childbearing potential should be advised to avoid becoming pregnant with an adequate method of contraception (barrier or hormonal methods) and men should be advised to not father a child while receiving treatment with azacytidine. All men and women of childbearing potential must use acceptable methods of birth control throughout the study as described below: Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment. Men should use adequate birth control for at least 30 days after the last administration of sorafenib. Post-menopausal women (defined as no menses for at least a year) and surgically sterilized women are not required to undergo a pregnancy test.
12. Females of childbearing potential Recommendation is for 2 effective contraceptive methods during the study. Adequate forms of contraception are double-barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral, depo provera, or injectable contraceptives, intrauterine devices, and tubal ligation.
13. Male patients with female partners who are of childbearing potential: Recommendation is for male and partner to use at least 2 effective contraceptive methods, as described above, during the study.
14. Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
15. INR less than 1.5. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.

Exclusion Criteria:

1. Nursing and pregnant females.
2. Patients with acute promyelocytic leukemia are excluded unless multiply refractory and no other standard treatment strategies are available to them
3. Patients with known allergy to sorafenib or azacitidine, mannitol or any of their components.
4. Patients with known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of sorafenib.
5. Patients with any other known disease (except carcinoma in-situ) or concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, cardiovascular disease including congestive heart failure, myocardial infarction within 6 months and poorly controlled hypertension, chronic renal disease (creatinine clearance < 20 ml/min using the Cockcroft and Gault formula)., or active uncontrolled infection) which could compromise participation in the study.
6. Patients with a known confirmed diagnosis of HIV infection or active viral hepatitis (B or C).
7. Patients who have had any major surgical procedure within 28 days of Day 1.
8. Patients unwilling or unable to comply with the protocol.
9. Patients with known malignant disease of the central nervous system or advanced malignant hepatic tumors.
10. Cardiac disease: Congestive heart failure greater than class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
11. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
12. Uncontrolled hypertension defined as systolic blood pressure greater than 140 mmHg or diastolic pressure greater than 90 mmHg, despite optimal medical management.
13. Active clinically serious infection greater than CTCAE v4. Grade 2 not controlled with antibiotics.
14. Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
15. Pulmonary hemorrhage/bleeding event greater than CTCAE v4. Grade 2 within 4 weeks of first dose of study drug.
16. Any other hemorrhage/bleeding event greater than CTCAE v4. Grade 3 within 4 weeks of first dose of study drug.
17. Serious non-healing wound, ulcer, or bone fracture.
18. Evidence or history of bleeding diathesis or coagulopathy
19. Known or suspected allergy to sorafenib or any agent given in the course of this trial.
20. Patients with a history of solid organ transplant
21. Patients with seizure disorder requiring medication (such as antiepileptics).
22. Use of strong CYP3A4 inducers (eg, St. John's wort, dexamethasone at a dose of greater than 16 mg daily, phenytoin, carbamazepine, rifabutin, phenobarbital, or rifampin within seven days of initiating dosing
23. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ohanian M, Garcia-Manero G, Levis M, Jabbour E, Daver N, Borthakur G, Kadia T, Pierce S, Burger J, Richie MA, Patel K, Andreeff M, Estrov Z, Cortes J, Kantarjian H, Ravandi F. Sorafenib Combined with 5-azacytidine in Older Patients with Untreated FLT3-ITD Mutated Acute Myeloid Leukemia. Am J Hematol. 2018 Sep;93(9):1136-1141. doi: 10.1002/ajh.25198. Epub 2018 Aug 31. PMID 30028037
- [Derived] Ravandi F, Alattar ML, Grunwald MR, Rudek MA, Rajkhowa T, Richie MA, Pierce S, Daver N, Garcia-Manero G, Faderl S, Nazha A, Konopleva M, Borthakur G, Burger J, Kadia T, Dellasala S, Andreeff M, Cortes J, Kantarjian H, Levis M. Phase 2 study of azacytidine plus sorafenib in patients with acute myeloid leukemia and FLT-3 internal tandem duplication mutation. Blood. 2013 Jun 6;121(23):4655-62. doi: 10.1182/blood-2013-01-480228. Epub 2013 Apr 23. PMID 23613521
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 11, 2011 to February 4, 2013. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Phase I: Azacitidine + Sorafenib: Azacitidine (AZA) 75 mg/m^2 subcutaneously (SQ) or intravenously (IV) daily for 7 days and Sorafenib starting dose 200 mg orally twice a day for 28 Day cycle.
- Phase II: Azacitidine + 400 mg Sorafenib: Azacitidine (AZA) 75 mg/m^2 subcutaneously (SQ) or intravenously (IV) daily for 7 days and Sorafenib 400 mg orally twice a day for 28 Day cycle.
Period: Overall Study
Arm/Group | Phase I: Azacitidine + Sorafenib | Phase II: Azacitidine + 400 mg Sorafenib
Started | 3 | 57
Completed | 2 | 47
Not Completed | 1 | 10
Not completed — Ineligible | 0 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Disease Progression | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Phase II: Azacitidine + 400 Sorafenib: Azacitidine (AZA) 75 mg/m^2 subcutaneously (SQ) or intravenously (IV) daily for 7 days and Sorafenib 400 mg orally twice a day for 28 Day cycle.
- Total: Total of all reporting groups
Arm/Group | Phase I: Azacitidine + Sorafenib | Phase II: Azacitidine + 400 Sorafenib | Total
Number analyzed (Participants) | 3 | 57 | 60
Age, Continuous [Median (Full Range); unit: years] | 73 [40 to 87] | 64 [20 to 81] | 64 [20 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 27 | 28
  Male | 2 | 30 | 32
Region of Enrollment [Number; unit: participants]
  United States | 3 | 57 | 60

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Sorafenib Given With Azacitidine
Description: MTD is defined as highest dose level in which 6 patients treated with at most 1 experiencing a dose limiting toxicity (DLT) during 1st cycle. One cycle of therapy is 7 days of azacitidine (AZA) and 28 days of sorafenib. Starting dose of Sorafenib is 200 mg twice a day azacitidine
Time Frame: 28 day cycle
Measure: Number; unit: mg/twice daily
Groups:
- Azacitidine + Sorafenib: Azacitidine (AZA) 75 mg/m^2 subcutaneously (SQ) or intravenously (IV) daily for 7 days and Sorafenib starting dose 200 mg orally twice a day for 28 Day cycle.
Arm/Group | Azacitidine + Sorafenib
Number analyzed (Participants) | 3
mg/twice daily | 400

2. Secondary Outcome: Phase II: Number of Participants With Response
Description: Response according to International Working Group response criteria for Acute myeloid leukemia (AML) (JCO 2003; 21: 4642-9): CR defined by presence of <5% blasts in the bone marrow (BM), with >1 X 10^9/L neutrophils and >100 x 10^9/L platelets in the peripheral blood (PB) with no detectable extramedullary disease. Participants who met the above criteria but had neutrophil or platelet counts less than the stated values were considered to have achieved CRi (CR with incomplete recovery of PB counts) or CR with incomplete platelet recovery (CRp) if CR but platelets < 100 x 10^9/L but ≥ 50 x 10^9/L and platelet transfusion independent. Partial response (PR) required all of the hematologic values for a CR but with a decrease of >/= 50% in the percentage of blasts to 5% to 25% in the BM aspirate.
Time Frame: 90 days
Population: Nine participants were not evaluable for response.
Measure: Number; unit: participants
Arm/Group | Azacitidine + Sorafenib
Number analyzed (Participants) | 48
participants
  Complete Response (CR) | 8
  Complete Remission Without Platelet Recovery (CRi) | 10
  Partial Response | 1
  Complete Response (CRp) | 6
  No Response | 23

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent to discontinuation of treatment, up to 1 year. Total study period was 3 years and 11 months.
Groups:
- Phase II: Azacitidine + Sorafenib: Azacitidine (AZA) 75 mg/m^2 subcutaneously (SQ) or intravenously (IV) daily for 7 days and Sorafenib starting dose 400 mg orally twice a day for 28 Day cycle.
Arm/Group | Phase I: Azacitidine + Sorafenib | Phase II: Azacitidine + Sorafenib
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/57
Other Adverse Events (participants affected / at risk) | 3/3 | 51/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Azacitidine + Sorafenib (N=3) | Phase II: Azacitidine + Sorafenib (N=57)
Alanine Aminotransferase (Metabolism and nutrition disorders) | 2 (2) | 19 (20)
Aspartate Aminotransferase (Metabolism and nutrition disorders) | 2 (2) | 22 (22)
Bilirubin (Metabolism and nutrition disorders) | 3 (3) | 28 (28)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 15 (15)
Fatigue (General disorders) | 2 (2) | 25 (25)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Irritability (Nervous system disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 12 (12)
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Metabolic/Lab (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Infections and infestations) | 1 (1) | 13 (14)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 14 (14)
Infection (documented clinically) (Infections and infestations) | 0 (0) | 26 (62)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (5)
Mucositis (clinical exam) (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 13 (13)
Neutrophils (Blood and lymphatic system disorders) | 0 (0) | 13 (13)
Pain (General disorders) | 0 (0) | 4 (4)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Hand-Foot (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Anorexia (Gastrointestinal disorders) | 0 (0) | 6 (6)
Infection with normal ANC (Infections and infestations) | 0 (0) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Weight Loss (General disorders) | 0 (0) | 4 (4)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Infection - Other (Infections and infestations) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 6 (6)
Mucositis (functional/symptomatic) (Gastrointestinal disorders) | 0 (0) | 3 (3)
Neuropathy - Sensory (Nervous system disorders) | 0 (0) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blurred Vision (Eye disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 1 (1)
Supraventricular Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac General-Other (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Infections and infestations) | 0 (0) | 1 (1)
Edema - Limb (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mental Status (Nervous system disorders) | 0 (0) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
CNS Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes